CLINICAL TRIAL: NCT01644890
Title: A Multi-national Phase III Clinical Study Comparing NK105 Versus Paclitaxel in Patients With Metastatic or Recurrent Breast Cancer
Brief Title: A Phase III Study of NK105 in Patients With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nippon Kayaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3105301
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2016-02

CONDITIONS: Breast Cancer Nos Metastatic Recurrent
Keywords: NK105, Paclitaxel, Breast cancer, Micelle
MeSH Terms: conditions — Breast Neoplasms | interventions — NK105; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NK105 (Experimental)
  Interventions: Drug: NK105
- Paclitaxel (Active Comparator)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: NK105 — IV, Weekly
  Arms: NK105
Drug: Paclitaxel — IV, Weekly
  Arms: Paclitaxel

SUMMARY:
To verify the non-inferiority of NK105, a paclitaxel-incorporating micellar nanoparticle, to paclitaxel in terms of the progression-free survival in patients with metastatic or recurrent breast cancer.

DETAILED DESCRIPTION:
This study is a randomized, open-label, multi-national phase III study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the patient signed by herself.
* Histologically confirmed metastatic or recurrent adenocarcinoma of the breast.
* Aged 20 to 74 at the time of informed consent.

Exclusion Criteria:

* Prior systemic chemotherapy with taxane anticancer drugs for metastatic or recurrent breast cancer.

Ages: 20 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2012-07; Primary Completion 2016-07 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call +81-3-6731-5200 Mon - Fri 9 AM - 5 PM (Japan Time), Study Director — Nippon Kayaku Co., Ltd.
Locations (1):
- Japan Sites, Tokyo, Etc., Japan

REFERENCES:
- [Derived] Fujiwara Y, Mukai H, Saeki T, Ro J, Lin YC, Nagai SE, Lee KS, Watanabe J, Ohtani S, Kim SB, Kuroi K, Tsugawa K, Tokuda Y, Iwata H, Park YH, Yang Y, Nambu Y. A multi-national, randomised, open-label, parallel, phase III non-inferiority study comparing NK105 and paclitaxel in metastatic or recurrent breast cancer patients. Br J Cancer. 2019 Mar;120(5):475-480. doi: 10.1038/s41416-019-0391-z. Epub 2019 Feb 12. PMID 30745582

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from September 2012 to January 2016 in three asian countries (Japan, Korea, Taiwan).
Groups:
- NK105: received NK105 (65 mg/m^2) on days 1, 8 and 15 of a 28-day cycle
- Paclitaxel: received Paclitaxel (80 mg/m^2) on days 1, 8 and 15 of a 28-day cycle
Period: Overall Study
Arm/Group | NK105 | Paclitaxel
Started | 218 | 218
Completed | 2 | 3
Not Completed | 216 | 215
Not completed — Adverse Event | 7 | 20
Not completed — Death | 1 | 3
Not completed — Physician Decision | 3 | 9
Not completed — Protocol Violation | 6 | 7
Not completed — Withdrawal by Subject | 19 | 27
Not completed — Progression Disease | 160 | 131
Not completed — Clinical Progression | 6 | 6
Not completed — > 28 days since last dose of study drug | 6 | 3
Not completed — Other | 8 | 9

BASELINE CHARACTERISTICS:
Population: All randomized patients who received study drug at least once
Groups:
- Total: Total of all reporting groups
Arm/Group | NK105 | Paclitaxel | Total
Number analyzed (Participants) | 214 | 213 | 427
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (10.3) | 55.0 (10.7) | 55.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214 | 213 | 427
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 136 | 143 | 279
  South Korea | 51 | 42 | 93
  Taiwan | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: PFS is defined as the period from the day of randomization until the first observation of lesion progression or death from any cause. Disease progression is defined as PD according to RECIST Ver. 1.1.
  Assessment period was from the day of randomisation until the first observation of lesion progression or death
Time Frame: Baseline, every 6 weeks of study treatment period, and end of study,
Population: All randomized patients who received study drug at least once and who had no major violations of the eligiblity criteria
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NK105 | Paclitaxel
Number analyzed (Participants) | 211 | 211
months | 8.4 [7.0 to 9.9] | 8.5 [6.9 to 11.5]
Statistical Analysis 1: Comparison: NK105 vs Paclitaxel; Based on the results of previous studies, the expected median PFS was 5.5 months for PTX and 6.35 months for NK105. Assuming a randomization period of 18 months, a follow-up period of 12 months, a one-sided significance level of 2.5%, a power of 85% and the non-inferiority margin of 1.215, the number of patients was estimated to 172 pts per group, a total of 344 patients. Considering an expected withdrawal/dropout rate of approximately 20%, the target sample size was set at 414; Test type: Non-Inferiority — The primary PFS analysis was confirmed whether or not the upper limit of the 95% confidence interval (CI) for the hazard ratio (HR) for NK105 relative to PTX fell below the non-inferiority margin of 1.215 (<1.215) by fitting a Cox proportional hazards model that included allocation adjustment factors other than the study site as covariates; Hazard Ratio (HR) = 1.255, 95% CI 2-sided [0.989 to 1.592] — History of chemotherapy for metastatic or recurrent breast cancer (yes/no), History of treatment using a taxane anticancer drug (yes/no), ER status [(+) or (-)], and Disease free interval (<12 months or ≥12 months) were covariates for adjustment

2. Secondary Outcome: Overall Survival
Description: OS is defined as the period from the day of randomization until the day of death from any cause.
  Assessment period was from the day of randomisation until the first observation of lesion progression or death
Time Frame: Baseline, every 6 weeks of study treatment period, and end of study.
Population: History of chemotherapy for metastatic or recurrent breast cancer (yes/no), History of treatment using a taxane anticancer drug (yes/no), ER status [ER (+) or ER (-)], and Disease free interval (<12 months or ≥12 months) were covariates for adjustment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NK105 | Paclitaxel
Number analyzed (Participants) | 211 | 211
months | 31.2 [27.1 to 39.3] | 36.2 [30.3 to NA] — NA = The upper limit of the Confidence Interval was not estimable as there were not enough events.
Statistical Analysis 1: Comparison: NK105 vs Paclitaxel; Test type: Other; Hazard Ratio (HR) = 1.197, 95% CI 2-sided [0.885 to 1.620] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Response Rate
Description: ORR is the proportion of patients who are assessed as complete response or partial response as the best overall response among evaluable patients, according to RECIST Ver.1.1.
  Assessment period was from the day of randomisation until the first observation of lesion progression or death
Time Frame: Baseline, every 6 weeks of study treatment period, and end of study.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | NK105 | Paclitaxel
Number analyzed (Participants) | 211 | 211
percentage of participants | 31.6 [25.0 to 38.7] | 39.0 [32.0 to 46.4]
Statistical Analysis 1: Comparison: NK105 vs Paclitaxel; Test type: Other; Difference in ORR (%) = -7.5, 95% CI 2-sided [-17.4 to 2.7]

ADVERSE EVENTS:
Time Frame: The duration of treatment, mean duration was 294.7 days.
Arm/Group | NK105 | Paclitaxel
All-Cause Mortality (participants affected / at risk) | 3/214 | 4/213
Serious Adverse Events (participants affected / at risk) | 34/214 | 27/213
Other Adverse Events (participants affected / at risk) | 210/214 | 211/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NK105 (N=214) | Paclitaxel (N=213)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Oesophageal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder perforation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NK105 (N=214) | Paclitaxel (N=211)
Anaemia (Blood and lymphatic system disorders) | 23 | 22
Abdominal pain upper (Gastrointestinal disorders) | 11 | 15
Constipation (Gastrointestinal disorders) | 37 | 42
Diarrhoea (Gastrointestinal disorders) | 47 | 41
Nausea (Gastrointestinal disorders) | 59 | 65
Stomatitis (Gastrointestinal disorders) | 42 | 46
Vomiting (Gastrointestinal disorders) | 31 | 25
Fatigue (General disorders) | 45 | 36
Influenza like illness (General disorders) | 5 | 12
Malaise (General disorders) | 21 | 37
Oedema (General disorders) | 6 | 23
Oedema peripheral (General disorders) | 15 | 41
Pyrexia (General disorders) | 22 | 27
Cystitis (Infections and infestations) | 11 | 13
Nasopharyngitis (Infections and infestations) | 49 | 46
Paronychia (Infections and infestations) | 7 | 16
Upper respiratory tract infection (Infections and infestations) | 26 | 25
Alanine aminotransferase increased (Investigations) | 24 | 22
Aspartate aminotransferase increased (Investigations) | 20 | 15
Gamma-glutamyltransferase increased (Investigations) | 20 | 14
Lymphocyte count decreased (Investigations) | 20 | 25
Neutrophil count decreased (Investigations) | 109 | 103
Weight decreased (Investigations) | 29 | 36
Weight increased (Investigations) | 22 | 26
White blood cell count decreased (Investigations) | 72 | 68
Decreased appetite (Metabolism and nutrition disorders) | 27 | 39
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 38
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 32 | 46
Dizziness (Nervous system disorders) | 12 | 20
Dysgeusia (Nervous system disorders) | 30 | 53
Headache (Nervous system disorders) | 29 | 36
Peripheral sensory neuropathy (Nervous system disorders) | 113 | 149
Insomnia (Psychiatric disorders) | 16 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 37 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 151 | 161
Nail discolouration (Skin and subcutaneous tissue disorders) | 37 | 46
Pruritus (Skin and subcutaneous tissue disorders) | 27 | 20
Rash (Skin and subcutaneous tissue disorders) | 62 | 47
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 17 | 12
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 11 | 5
Onychomadesis (Skin and subcutaneous tissue disorders) | 4 | 15
Hot flush (Vascular disorders) | 4 | 12

LIMITATIONS AND CAVEATS:
No limitation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is no day limit but it needs sponsor's consent in a document.